CLINICAL TRIAL: NCT02156544
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Single Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of CKD-519 After Oral Administration in Healthy Adult Volunteers
Brief Title: Study to Investigate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of CKD-519
Acronym: CKD-519 FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 148HPS14001
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2014-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — CKD-519

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CKD-519 25mg (Experimental): CKD-519 25mg or placebo
  Interventions: Drug: CKD-519; Drug: placebo
- CKD-519 50mg (Experimental): CKD-519 50mg or placebo
  Interventions: Drug: CKD-519; Drug: placebo
- CKD-519 100mg (Experimental): CKD-519 100mg or placebo
  Interventions: Drug: CKD-519; Drug: placebo
- CKD-519 200mg (Experimental): CKD-519 200mg or placebo
  Interventions: Drug: CKD-519; Drug: placebo
- CKD-519 400mg (Experimental): CKD-519 400mg or placebo
  Interventions: Drug: CKD-519; Drug: placebo

INTERVENTIONS:
Drug: CKD-519
Drug: placebo

SUMMARY:
The purpose of this study is to investigate the safety/tolerability and pharmacokinetics/pharmacodynamics of CKD-519.

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 55 aged in healthy adult
2. Body weight more than 55kg in male, 50kg in female
3. Body Mass Index more than 18.5 and under 25(body mass index=kg/m2)
4. If female, must include more than one among the items

   * The menopause(there is no natural menses for at least 2 years)
   * Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition
5. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms and do not sperm donation until two months during clinical trials and after the final dosage of investigational products
6. Those who fully understand about this clinical trials after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system(severe hepatic impairment, etc), kidney(severe renal impairment, etc), nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system(heart failure, etc) or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption(Crohn's disease, ulcers, etc.) or surgery(except simple appendectomy or hernia surgery)
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of drugs or additives.
4. An impossible one who participates in clinical trial including screening tests(medical history taking, BP, 12-lead ECG, physical examination, blood&urine laboratory test result) before 28 days the taking investigational Products.
5. Defined by the following laboratory parameters

   * AST, ALT>1.25* upper limit of normal range
   * Total bilirubin>1.5* upper limit of normal range
   * CPK>1.5* upper limit of normal range
   * eGFR(using by MDRD method)<60mL/min/1.73m2
6. Sitting SBP>150mmHg or <90mmHg, sitting DBP>100mmHg or <50mmHg, after 5 minutes break.
7. Drug abuse or have a history of drug abuse showes a positive for urine drug test.
8. Pregnant or lactating women.
9. A heavy caffeine consumer(caffeine>5 cups/day), alcohol consumer(alcohol>210g/week), or smoker(cigarette>10 cigarettes/day)
10. Subject takes ethical drug or herbal medicine within 14 days, OTC within 7 days before the beginning of study treatment but investigator determine that the taking drug affect this study or could affect the safety of subjects.
11. Subject who takes inhibitor and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30 days.
12. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1L per a day or more within 7 days before the beginning of study treatment)
13. Subject who treated with any investigational drugs within 60 days before the beginning of study treatment(However, biologicals applies for 90 days, but can be based on a more extended period of time by considering the half-life)
14. Previously donate whole blood within 60 days or component blood within 30 days.
15. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
16. Positive for Serology test(Hepatitis B, Hepatitis C, HIV)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-519 | 0(predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
AUC0-last of CKD-519 | 0(predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
AUC0-∞ of CKD-519 | 0(Predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
Tmax of CKD-519 | 0(Predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
t1/2 of CKD-519 | 0(Predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
CL/F of CKD-519 | 0(Predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
Vd/F of CKD-519 | 0(Predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168

SECONDARY OUTCOMES:
CETP activity | 0(Predose), 0.5, 1, 2, 4, 8, 18, 24, 48, 72, 96, 120, 144, 168

CONTACTS AND LOCATIONS:
Overall Officials: Min-Su Park, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea